CLINICAL TRIAL: NCT05765994
Title: The Effects of Small Intestinal Bacterial Overgrowth Syndrome in ICU Patients. An Observational Study
Brief Title: Small Intestinal Bacterial Overgrowth in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Agathi Karakosta, Assistant Professor of Anaesthesiology, University of Ioannina
Other Study IDs: 207
Record Dates: First submitted 2023-02-25; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Small Intestinal Bacterial Overgrowth; Critical Illness; Intensive Care Unit
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients: Adult ICU patients on mechanical ventilation
  Interventions: Diagnostic Test: Modified hydrogen breath test

INTERVENTIONS:
Diagnostic Test: Modified hydrogen breath test — A modified technique to obtain expired hydrogen from the ventilator tubes is performed. A connection with a valve attached to a collecting bag is inserted at the end of the expiratory limb of the breathing circuit for exhaled air collection.
  Other Names: Hydrogen monitor Gastrolyzer / Gastro+TM (Bedfont® Scientific Ltd,) was used for expired hydrogen (eH2) testing.

SUMMARY:
Small intestinal bacterial overgrowth (SIBO) syndrome, though associated with potentially serious complications, has not been adequately studied to date in critically ill patients hospitalized in intensive care units (ICU).

A modified method for SIBO diagnosis is employed concerning a standard breath test. Specifically, as all participants are intubated and in need of mechanical ventilation, SIBO diagnosis is based on a non-invasive modified technique for sampling exhaled air from the ventilator tubes and performing a standard hydrogen breath test.

The primary objective of this study is assessment of the prevalence of SIBO on ICU patients. Secondary outcomes include investigation of the effects of SIBO on ventilator associated pneumonia, as well as ICU length of stay and all-cause in-hospital mortality rate in critically ill patients.

DETAILED DESCRIPTION:
Small intestine bacterial overgrowth (SIBO) remains to this day a syndrome that is not fully understood. Initially, it was considered quite rare, but today there are reports suggesting a SIBO prevalence between 6 to 15% of healthy, asymptomatic people and reaching 80% in patients with irritable bowel syndrome. It is often involved in various disorders, such as diarrhea and malabsorption. It is defined as an increase in the number and/or disturbance in the type of bacteria in the upper part of the intestinal tract.

SIBO occurs when the homeostatic mechanisms of the small intestine are disturbed. The two main conditions that favor microbial overgrowth in the small intestine are decreased acid secretion from the stomach and small bowel dyskinesia.

The literature is scarce concerning the effects of SIBO on critically ill patients. To our knowledge this is the first study investigating the effects of SIBO on mechanically ventilated patients. It is a non-invasive observational study employing a modified technique to obtain exhaled air from the ventilator tubes to perform a standard hydrogen breath test for SIBO diagnosis. Lactulose is used as a substrate. Specifically, each patient is administered 20 g of lactulose diluted in 400 ml of water through the nasogastric tube. Measurements are performed at 0-15-30-45-60-90-120-180 min from lactulose administration. During measurements, a valve attached to a collecting bag at the end of the expiratory limb of the breathing circuit, is kept open and the collecting bag is filled by several patient exhalations. After valve closure and bag isolation, the air is drawn by a 50 ml polyethylene syringe which is connected to the valve system to prevent losses and/or contamination. Then the air is blown into the breath hydrogen monitor and the expired hydrogen measurement is recorded.

The hydrogen breath test is repeated at predetermined, protocol-based time intervals for all participants included in the study; 1st/day of admission, 3rd, 5th and 7th day of ICU stay. The 1st day measurement serves as a measure of eligibility, and patients exhibiting abnormal values of hydrogen breath testing at Day 1 are excluded from the study.

An increase by more than 20 ppm of eH2 from baseline within 90 min was considered an abnormal measurement suggesting SIBO. Moreover, an increase by more than 12 ppm of eH2 from baseline within the first 30 minutes followed by a second rise within the next 15 minutes (double peak) was also considered an abnormal measurement suggesting SIBO.

The primary objective of this study is assessment of the prevalence of SIBO on critically ill mechanically ventilated ICU patients. Secondary outcomes include investigation of the effects of SIBO on ventilator associated pneumonia, as well as ICU length of stay and all-cause in-hospital mortality rate in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients, in need of mechanical ventilation with an expected ICU length of stay and expected mechanical ventilation duration of more than 48 hours

Exclusion Criteria:

* abnormal hydrogen breath test on the day of ICU admission (Day 1)
* recent (up to four weeks before ICU admission) antimicrobial therapy or patients already receiving antimicrobial therapy on admission
* recent (up to four weeks before ICU admission) use of gastroprotective medication, probiotics and prokinetics
* patients with known gastrointestinal disease prior to admission
* recent abdominal surgery resulting in planned or unplanned ICU admission
* extubation or death before protocol completion (7 days) constitute exclusion criteria after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients admitted to the ICU and in need of mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
SIBO prevalence | From date of ICU admission to date of ICU discharge or date of death from any cause, whichever came first, assessed up to one month)
  The proportion of ICU patients diagnosed with SIBO

SECONDARY OUTCOMES:
VAP (ventilator associated pneumonia) | From date of ICU admission to date of ICU discharge or date of death from any cause, whichever came first, assessed up to one month)
  The proportion of ICU patients diagnosed with VAP
ICU LOS | From date of ICU admission to date of ICU discharge or date of death from any cause, whichever came first, assessed up to one month)
  ICU lenght of stay, days
All-cause in-hospital mortality | From date of ICU admission to date of ICU discharge or date of death from any cause, whichever came first, assessed up to one month)
  Death due to any cause during ICU and hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Univesity Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Undecided